CLINICAL TRIAL: NCT02988271
Title: Self-Administered Meditation Intervention for Cancer Patients With Psychosocial Distress
Brief Title: Meditation Therapy in Improving Anxiety and Depression in Cancer Patients With Psychosocial Distress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0491; NCI-2018-01295 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0491 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Malignant Neoplasm
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms | interventions — Interviews as Topic; Meditation; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (meditation) (Experimental): Patients watch a pre-recorded instructional meditation video via an iPod meditation app. Patients then complete meditation exercises using the meditation app over 5-15 minutes QD for up to 2 weeks. Patients also complete questionnaires before and after meditation sessions and participate in an interview over 10 minutes.
  Interventions: Other: Interview; Procedure: Meditation Therapy; Procedure: Quality-of-Life Assessment
- Group II (waitlist control) (Active Comparator): Patients receive supportive care, such as access to social workers, support groups, spiritual care, or other patient services for up to 2 weeks. Patients also complete questionnaires over 15-20 minutes and participate in an interview over 10 minutes.
  Interventions: Other: Interview; Procedure: Quality-of-Life Assessment; Procedure: Supportive Care

INTERVENTIONS:
Other: Interview — Participate in interview
Procedure: Meditation Therapy — Complete meditation therapy
  Other Names: Meditation
  Arms: Group I (meditation)
Procedure: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Procedure: Supportive Care — Receive supportive care
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Group II (waitlist control)

SUMMARY:
This trial studies how well self-administered meditation therapy works in improving anxiety and depression in cancer patients who exhibit psychosocial distress. Meditation therapy is a mind-body approach that uses a variety of techniques, such as deep breathing, sound, or movement, that may help to decrease distress and anxiety and enhance the health and quality of life of patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of having patients self-administer meditation recordings using a portable, computer-based program during a 2-week period.

SECONDARY OBJECTIVES:

I. Assess the effect of self-administered meditation on anxiety, depression and other symptoms that are part of the Edmonton Symptom Assessment Scale (ESAS) questionnaire.

II. Evaluate participant satisfaction with the meditation delivery and tracking program.

III. Examine the association between the frequency of practice (number of sessions a day) and choice of length of practice (5, 10, or 15 minute sessions) and anxiety, depression and other patient reported outcomes.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (MEDITATION): Patients watch a pre-recorded instructional meditation video via an iPod meditation app. Patients then complete meditation exercises using the meditation app over 5-15 minutes once daily (QD) for up to 2 weeks. Patients also complete questionnaires before and after meditation sessions and participate in an interview over 10 minutes.

GROUP II (WAITLIST CONTROL): Patients receive supportive care, such as access to social workers, support groups, spiritual care, or other patient services for up to 2 weeks. Patients also complete questionnaires over 15-20 minutes and participate in an interview over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients at MD Anderson with a cancer history who are either undergoing active treatment or who have completed treatment for their cancer
* Must understand and read English, sign a written informed consent, and follow protocol requirements
* Willing to come to MD Anderson Main Campus (Texas Medical Center) for enrollment
* Patient self-reported ESAS psychological scale score (sum of anxiety and depression scores) between 4 and 11 (and/or) individual anxiety or depression score between 4 and 7 on a 0 to 10 numeric scale, where 10 is the worst possible
* If on medication for anxiety, stable dose of medications for management of anxiety symptoms for at least six weeks prior to enrollment with no plans to change meditations in the subsequent four weeks. Increases or decreases allowed within drug class, but changing drug class will make patient in-evaluable

Exclusion Criteria:

* Diagnosis of a formal thought disorder (e.g., schizophrenia)
* Known history of a neurological and/or psychological disorder that in the physician's opinion may interfere with the patient's ability to cooperate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of self-administered meditation | Up to 2 weeks
  Feasibility will be confirmed if at least 50% of the eligible patients approached consent to the study and at least 70% of subjects complete at least two meditation sessions each week during the 2-week period. The study will calculate rates, frequencies, and 90% confidence intervals (CIs) of the rates.

SECONDARY OUTCOMES:
Self-administered meditation effect on anxiety and depression as measured by the Edmonton Symptom Assessment Scale (ESAS) questionnaire | Up to 2 weeks
  Summary statistics and 90% CIs will be calculated to assess differences in mean anxiety, depression and other outcomes measured at the end of the study, as well as the change scores from baseline, between subjects randomized to meditation and those randomized to wait-list. Additional analysis may include analysis of covariance (ANCOVA) to control for relevant baseline outcome variables or other patient characteristics. Summary statistics and 90% CIs will also be calculated separately by intervention arm and to examine within-subject differences for those who were randomized to wait-list and then received the meditation intervention.
The study will evaluate participant satisfaction with the meditation delivery and tracking program using appropriate descriptive statistics. | Up to 2 weeks
  The questionnaire purpose is to learn more about meditation's effect on your health over the past two weeks. It asks, how much do you agree or disagree? Options are, strongly disagree, disagree, neutral, agree and strongly agree. The questionnaire asks patients to pick the closest answer for each statement. The first statements asks, 'My well-being has improved', the second, "I am more focused', the third asks, 'I am in a better mood', the fourth asks, 'My energy level had increased', and lastly, 'I am sleeping better'. The exit questionnaire is scored as a sum value for each scale range provided. For each scale range provided, higher values/and or lower values represent whether participants agree or disagree with the statements listed.
Frequency of meditation and choice of length of meditation | Up to 2 weeks
  The study will explore the association between frequency of meditation and choice of length of meditation and patient reported outcomes using correlation analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Lopez, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org